CLINICAL TRIAL: NCT02158546
Title: A Phase 3 Efficacy and Safety Study of ALKS 5461 for the Adjunctive Treatment of Major Depressive Disorder (the FORWARD-3 Study)
Brief Title: A Study of ALKS 5461 for the Treatment of Major Depressive Disorder (MDD) - the FORWARD-3 Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alkermes, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ALK5461-206
Record Dates: First submitted 2014-06-05; First posted 2014-06-09 (Estimated); Results first posted 2019-06-25 (Actual); Last update posted 2019-06-25 (Actual); Status verified 2019-05

CONDITIONS: Major Depressive Disorder
Keywords: Major Depressive Disorder; Depression; Alkermes; ALKS 5461; Samidorphan
MeSH Terms: conditions — Depressive Disorder, Major; Depression | interventions — ALKS 5461

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- ALKS 5461 (Experimental)
  Interventions: Drug: ALKS 5461
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ALKS 5461 — Sublingual tablet, taken once daily (in addition to open-label treatment with a commercially available antidepressant)
  Arms: ALKS 5461
Drug: Placebo — Sublingual tablet, taken once daily (in addition to open-label treatment with a commercially available antidepressant)
  Arms: Placebo

SUMMARY:
This study will evaluate the efficacy and safety of ALKS 5461.

ELIGIBILITY:
Inclusion Criteria:

* Have a Body Mass Index (BMI) of 18.0 to 40.0 kg/m2, inclusive
* Agree to use an acceptable method of contraception for the duration of the study
* Have a Major Depressive Disorder (MDD) primary diagnosis
* Have no more than 2 inadequate responses to antidepressant therapy (ADT) in the current Major Depressive Episode (MDE)
* Additional criteria may apply

Exclusion Criteria:

* Have a current primary Axis-I disorder other than MDD
* Have used opioid agonists (eg, codeine, oxycodone, tramadol, morphine) or opioid antagonists (eg, naloxone, naltrexone) within 14 days
* Have received electroconvulsive therapy treatment within the last 2 years or received more than one course of electroconvulsive treatment during lifetime
* Have attempted suicide within the past 2 years
* Have a positive test for drugs of abuse
* Are pregnant, planning to become pregnant, or breastfeeding
* Have a history of intolerance, allergy, or hypersensitivity to buprenorphine or opioid antagonists (eg, naltrexone, naloxone)
* Have had a significant blood loss or blood donation within 60 days
* Additional criteria may apply

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 447 (Actual)
Dates: Start 2014-05; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sanjeev Pathak, MD, Study Director — Alkermes, Inc.
Locations (54):
- United States (48):
  - Alkermes Investigational Site, Little Rock, Arkansas
  - Alkermes Investigational Site, Bellflower, California
  - Alkermes Investigational Site, Beverly Hills, California
  - Alkermes Investigational Site, Glendale, California
  - Alkermes Investigational Site, Los Alamitos, California
  - Alkermes Investigational Site, Orange, California
  - Alkermes Investigational Site, Redlands, California
  - Alkermes Investigational Site, Temecula, California
  - Alkermes Investigational Site, Washington D.C., District of Columbia
  - Alkermes Investigational Site, Hallandale, Florida
  - Alkermes Investigational Site, Hialeah, Florida
  - Alkermes Investigational Site, Jacksonville, Florida
  - Alkermes Investigational Site, Leesburg, Florida
  - Alkermes Investigational Site, Maitland, Florida
  - Alkermes Investigational Site, Tampa, Florida
  - Alkermes Investigational Site, Atlanta, Georgia
  - Alkermes Investigational Site, Chicago, Illinois
  - Alkermes Investigational Site, Oak Brook, Illinois
  - Alkermes Investigational Site, Vernon Hills, Illinois
  - Alkermes Investigational Site, Indianapolis, Indiana
  - Alkermes Investigational Site, Lafayette, Indiana
  - Alkermes Investigational Site, Edgewood, Kentucky
  - Alkermes Investigational, Washington DC, Maryland
  - Alkermes Investigational Site, Brockton, Massachusetts
  - Alkermes Investigational Site, Watertown, Massachusetts
  - Alkermes Investigational Site, Kansas City, Missouri
  - Alkermes Investigational Site, O'Fallon, Missouri
  - Alkermes Investigational Site, St Louis, Missouri
  - Alkermes Investigational Site, Cherry Hill, New Jersey
  - Alkermes Investigational Site, Albuquerque, New Mexico
  - Alkermes Investigational Site, Jamaica, New York
  - Alkermes Investigational Site, New York, New York
  - Alkermes Investigational Site, Staten Island, New York
  - Alkermes Investigational Site, Charlotte, North Carolina
  - Alkermes Investigational Site, Beachwood, Ohio
  - Alkermes Investigational Site, Cincinnati, Ohio
  - Alkermes Investigational Site, Mason, Ohio
  - Alkermes Investigational Site, Middleburg Heights, Ohio
  - Alkermes Investigational Site, Portland, Oregon
  - Alkermes Investigational Site, Salem, Oregon
  - Alkermes Investigational Site, Philadelphia, Pennsylvania
  - Alkermes Investigational Site, Charleston, South Carolina
  - Alkermes Investigational Site, Memphis, Tennessee
  - Alkermes Investigational Site, Dallas, Texas
  - Alkermes Investigational Site, Houston, Texas
  - Alkermes Investigational Site, Sugar Land, Texas
  - Alkermes Investigational Site, Bellevue, Washington
  - Alkermes Investigational Site, Waukesha, Wisconsin
- Bulgaria (6):
  - Alkermes Investigational Site, Burgas
  - Alkermes Investigational Site, Kazanlak
  - Alkermes Investigational Site, Sofia
  - Alkermes Investigational Site, Varna
  - Alkermes Investigational Site, Veliko Tarnovo
  - Alkermes Investigational Site, Vratsa

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were diagnosed with major depressive disorder (MDD) and had an inadequate response to 1 or 2 adequate courses of treatment with a commercially available antidepressant therapy (ADT) during the current major depressive episode (MDE). All subjects continued ADT for the duration of the study.
Pre-assignment Details: 2 cohorts of subjects were enrolled: Group 1- subjects with baseline HAM-D17 score ≥ 20; Group 2- subjects with baseline HAM-D17 score 18-19. Only Group 1 was included in the efficacy analysis. Study included a 4-week pbo run-in period prior to the 6-week treatment period. In Group 1, 102 subjects did not meet criteria for randomization.
Groups:
- Group 1 - ALKS 5461 2mg/2mg; Group 2 ALKS 5461 2mg/2mg: Randomized to ALKS 5461 2mg/2mg
- Group 1 - Placebo; Group 2 - Placebo: Randomized to Placebo
Period: Overall Study
Arm/Group | Group 1 - ALKS 5461 2mg/2mg | Group 1 - Placebo | Group 2 ALKS 5461 2mg/2mg | Group 2 - Placebo
Started (3 subjects were randomized but did not receive study drug.) | 152 | 153 | 18 | 19
Completed | 133 | 136 | 14 | 13
Not Completed | 19 | 17 | 4 | 6
Not completed — Physician Decision | 0 | 1 | 0 | 0
Not completed — Non-compliance | 0 | 1 | 0 | 1
Not completed — Failure to meet eligibility criteria | 0 | 1 | 0 | 0
Not completed — Lack of Efficacy | 1 | 1 | 0 | 0
Not completed — Adverse Event | 2 | 2 | 0 | 0
Not completed — Withdrawal by Subject | 6 | 2 | 1 | 0
Not completed — Lost to Follow-up | 5 | 4 | 0 | 1
Not completed — Site Excluded | 5 | 5 | 3 | 4

BASELINE CHARACTERISTICS:
Population: Baseline data is presented for all subjects randomized to treatment. Data from 1 site (18 subjects) was excluded due to data integrity concerns.
Groups:
- Group 1 ALKS 5461 2mg/2mg; Group 2 ALKS 5461 2mg/2mg: Randomized to ALKS 5461 2mg/2mg
- Group 1 Placebo; Group 2 Placebo: Randomized to placebo
- Total: Total of all reporting groups
Arm/Group | Group 1 ALKS 5461 2mg/2mg | Group 1 Placebo | Group 2 ALKS 5461 2mg/2mg | Group 2 Placebo | Total
Number analyzed (Participants) | 147 | 148 | 15 | 15 | 325
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.4 (12.31) | 48.1 (12.51) | 47.5 (12.63) | 45.9 (11.44) | 47.7 (12.33)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 88 | 94 | 8 | 7 | 197
  Male | 59 | 54 | 7 | 8 | 128
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 23 | 29 | 2 | 1 | 55
  Not Hispanic or Latino | 124 | 119 | 13 | 14 | 270
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 0 | 0 | 0 | 2
  Asian | 5 | 0 | 0 | 0 | 5
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 0 | 0 | 1
  Black or African American | 33 | 33 | 3 | 2 | 71
  White | 106 | 115 | 12 | 13 | 246
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 118 | 128 | 14 | 12 | 272
  Bulgaria | 29 | 20 | 1 | 3 | 53

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to End of Treatment (Week 6) in the Montgomery Asberg Depression Rating Scale (MADRS) Total Score
Description: The MADRS-10 scale is a clinician-administered questionnaire comprised of 10 items used to measure the severity of MDD symptoms. Scores range from 0 (no apparent symptoms) to 60 (most severe symptoms). Individual questionnaire items include: Apparent Sadness, Reported Sadness, Inner Tension, Reduced Sleep, Reduced Appetite, Concentration Difficulties, Lassitude, Inability to Feel, Pessimistic Thoughts, and Suicidal Thoughts.
Time Frame: Baseline and week 6
Population: The Full Analysis Set (FAS) consists of subjects in the Group 1 Safety Population who have at least 1 post-randomization assessment of MADRS total score.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Groups:
- ALKS 5461 2mg/2mg: Randomized to ALKS 5461 2mg/2mg
- Placebo: Randomized to placebo
Arm/Group | ALKS 5461 2mg/2mg | Placebo
Number analyzed (Participants) | 142 | 146
units on a scale | -4.8 (0.67) | -4.6 (0.66)
Statistical Analysis 1: Comparison: ALKS 5461 2mg/2mg vs Placebo; Test type: Superiority; p = 0.782, Mixed Models Analysis; Least square means difference = -0.3, 95% CI 2-sided [-2.1 to 1.6], Standard Error of Mean 0.95

2. Secondary Outcome: Proportion of Patients Who Exhibited Treatment Response (MADRS-10)
Description: The proportion of subjects demonstrating MADRS-10 treatment response, defined as a ≥ 50% reduction in MADRS-10 score from baseline to the end of the efficacy period (week 6).
Time Frame: 6 weeks
Population: The FAS consists of subjects in the Group 1 Safety Population who have at least 1 post-randomization assessment of MADRS total score.
Measure: Count of Participants; unit: Participants
Arm/Group | ALKS 5461 2mg/2mg | Placebo
Number analyzed (Participants) | 142 | 146
Participants | 24 | 21

3. Secondary Outcome: Remission Rate
Description: The proportion of subjects achieving remission, defined as a MADRS-10 score of ≤ 10 at the end of the efficacy period.
Time Frame: 6 weeks
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | ALKS 5461 2mg/2mg | Placebo
Number analyzed (Participants) | 142 | 146
Participants | 20 | 18

4. Secondary Outcome: Number of Subjects With Adverse Events (AEs)
Time Frame: 6 weeks
Population: Safety population consisted of subjects who were identified as placebo non-responders at the end of the double-blind placebo run-in period and received at least one dose of randomized study drug (ie, placebo or ALKS 5461) subsequent to randomization.
Measure: Count of Participants; unit: Participants
Arm/Group | ALKS 5461 2mg/2mg | Placebo | Group 2 ALKS 5461 2mg/2mg | Group 2 Placebo
Number analyzed (Participants) | 147 | 148 | 15 | 15
Participants | 63 | 51 | 11 | 8

ADVERSE EVENTS:
Time Frame: AE reporting includes the 6-week double-blind, placebo-controlled period.
Arm/Group | Group 1 ALKS 5461 2mg/2mg | Group 1 Placebo | Group 2 ALKS 5461 2mg/2mg | Group 2 Placebo
All-Cause Mortality (participants affected / at risk) | 0/147 | 0/148 | 0/15 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/147 | 1/148 | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 39/147 | 24/148 | 11/15 | 8/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1 ALKS 5461 2mg/2mg (N=147) | Group 1 Placebo (N=148) | Group 2 ALKS 5461 2mg/2mg (N=15) | Group 2 Placebo (N=15)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1 ALKS 5461 2mg/2mg (N=147) | Group 1 Placebo (N=148) | Group 2 ALKS 5461 2mg/2mg (N=15) | Group 2 Placebo (N=15)
Nausea (Gastrointestinal disorders) | 13 (14) | 1 (1) | 4 (7) | 2 (2)
Vomiting (Gastrointestinal disorders) | 4 (4) | 2 (2) | 1 (2) | 0 (0)
Constipation (Gastrointestinal disorders) | 3 (3) | 1 (1) | 3 (3) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 3 (3) | 2 (2) | 2 (2) | 1 (1)
Fatigue (General disorders) | 4 (4) | 3 (3) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 4 (5) | 3 (4) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 3 (3) | 3 (3) | 0 (0) | 1 (1)
Blood creatine phosphokinase increased (Investigations) | 4 (4) | 0 (0) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 6 (7) | 5 (7) | 4 (4) | 1 (1)
Hypertension (Vascular disorders) | 3 (3) | 2 (2) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 3 (3) | 1 (2) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 3 (3) | 2 (2) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Eyelid oedema (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Food poisoning (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gingival pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Epicondylitis (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tooth fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood pressure increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urine output increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Metabolic syndorome (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Burning sensation (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Disturbance in attention (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypersomnia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Memory impairment (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Tension headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abnormal dreams (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nightmare (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sleep disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Initial insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Pre-specified primary population data are shown. Data from one trial site were excluded as pre-specified due to data integrity concerns (18 subjects). Other excluded subjects did not receive randomized study drug.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Should an Investigator desire to disclose study results, Sponsor will review the results disclosure prior to public release and can embargo the disclosure for a period of at least 60 days. Revisions to the disclosure will be negotiated in good faith. For a multicenter study the Investigators agree to publish/publicly present the results together with the other sites for the 12 month period after study results are available unless Sponsor grants written permission in advance.